CLINICAL TRIAL: NCT00209391
Title: A Multicentre, Phase 3, Open-Label, Controlled Study Evaluating the Efficacy and Safety of 0.1 mmol/kg OMNISCAN (Gadodiamide Injection) in Magnetic Resonance Angiography (MRA) of the Renal Arteries
Brief Title: A Safety & Efficacy Clinical Study to Evaluate the Narrowing of the Renal Arteries While Using Gadodiamide
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SOV301
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Renal Artery Stenosis
Keywords: Renal Artery Stenosis; Occlusion; Diagnostic Imaging; Omniscan; Magnetic Resonance Angiography; Contrast Media
MeSH Terms: conditions — Renal Artery Obstruction; Bites and Stings | interventions — gadodiamide

STUDY DESIGN:
Oversight: FDA-regulated Device: No

ARMS (1):
- Gadodiamide Injection (Experimental): All subjects will receive a single intravenous bolus injection via a power injector of Omniscan (Gadodiamide injection) at a dose of 0.1 mmol/kg.
  Interventions: Drug: Gadodiamide Injection

INTERVENTIONS:
Drug: Gadodiamide Injection
  Other Names: Omniscan

SUMMARY:
Magnetic Resonance Angiography (MRA) is an examination similar to Magnetic Resonance Imaging (MRI) which uses a magnetic field and a contrast medium when needed to visualize blood flow in the arterial vessels throughout the body.

Gadodiamide, a contrast medium, is already approved and is used to image blood vessels by directly injecting it into the vein, but this procedure has not been formally tested to image the renal artery vessels using MR.

The study is designed to determine the presence or absence of a relevant stenosis (ie greater than/equal to 50%) or occlusion in renal arteries. Intra-arterial Digital Subtraction Angiography will be used as the standard of truth.

DETAILED DESCRIPTION:
GEHC has decided not to provide this detail.

ELIGIBILITY:
Inclusion Criteria:

* Study Subjects must be adults with confirmed or suspected Renal Artery stenosis.
* The subject must have been referred for Digital Subtraction Angiography.

Exclusion Criteria:

* The subject has a known hypersensitivity to either conventional X-ray or gadolinium-based MR contrast media including, but not restricted to, the investigational product.
* The subject is lactating.
* The subject is pregnant as defined by a serum or urine β-HCG pregnancy test obtained within 24 hours before investigational product administration.
* The subject has received or is scheduled to receive MRI contrast medium within 24 h prior to or less than 24 hours after the investigational product administration.
* The subject has received or is scheduled to receive X-ray contrast medium within 7 days prior to or less than 24 hours after administration of investigational product.
* The subject has received an investigational product within 30 days prior to or will receive an investigational product less than 24 hours after investigational product administration.
* The subject has an active, serious, life-threatening disease with a life expectancy of less than 6 months.
* The subject has had a percutaneous transluminal angioplasty (PTA) in the renal region performed within 4 weeks prior to investigational product administration.
* The subject has a stent in the renal arteries.
* The subject has had a kidney transplantation.
* The subject has a serum creatinine value of >3.5 mg/dL (309.4 µmol/L).
* The subject has previously been included in this study.
* The subject has a contra-indication for MRI according to accepted clinical guidelines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2003-09; Primary Completion 2005-08-01 (Actual); Study Completion 2005-08-01 (Actual)

PRIMARY OUTCOMES:
Subject level efficacy of CE-MRA in detecting stenosis (50% occlusion) of major renal arteries. IA-DSA is the truth standard. | 72 hours

SECONDARY OUTCOMES:
Subject and vessel level efficacy comparison of CE-MRA and TOF-MRA in detecting stenosis, accessing arteries and diagnosis; Efficacy of CE-MRA and TOF-MAR combined; Clinical utility; Safety | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Michael Karl, PhD, Study Director — GE Healthcare
Locations (1):
- Amersham Buchler GmbH & Co. KG, Ismaning, Germany